CLINICAL TRIAL: NCT03176914
Title: Testing the Effectiveness of a Modified Care Group Model in Improving Child Health Outcomes in Mashonaland East, Zimbabwe
Brief Title: Testing the Effectiveness of a Modified Community Model in Improving Child Health Outcomes in Mashonaland East, Zimbabwe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zimbabwe (Other)
Collaborators: NORHED (Unknown)
Responsible Party: Principal Investigator, Maxwell Mhlanga, Principal Investigator, University of Zimbabwe
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MRCZ/A/2099
Record Dates: First submitted 2017-05-24; First posted 2017-06-06 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Pneumonia; Diarrhea; Malnutrition; Fever
Keywords: Community mobilisation
MeSH Terms: conditions — Pneumonia; Diarrhea; Malnutrition; Fever

STUDY DESIGN:
Intervention Model Description: The study will have an intervention arm under which the study intervention will be implemented and this will be compared with the outcomes in the conventional intervention arm. Each arm will have 11 clusters of an average size of 50.
Who Masked: Outcomes Assessor
Masking Description: The data analysts will be provided with coded data that doesn't reflect which arm the data is from.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Eleven clusters (Villages) will be randomly selected. A cluster will comprises of 10-15 volunteers selected from a cohort 10-15 households. Educative sessions will be held in each cluster once every fortnight using a participatory methods by a trained Village Health Worker (VHW). A session will focus on one thematic area running for 1-2 hours. Trained volunteers will in turn replicate the session(s) in their cohorts and do home visits to monitor care practices and screen children for various ailment. Health information is collated from each cluster and consolidated by the VHW who reports monthly at the clinic.
  Interventions: Behavioral: prevention and management of childhood illnesses at community level
- Conventional Intervention arm (Active Comparator): In the conventional mobilization system, a Village Health Worker facilitates community health programs as the sole source of health education for the entire villages. She does home visits, child growth monitoring and the various components primary health care at village level inclusive of disease surveillance and community case management using the 'supermarket approach' , whereby 3 or more themes are covered in a space of 10- 30 minutes in functions like funerals, village gatherings and other opportune moments. The Village Health worker prepares village monthly reports on all the indicators on community health and submits to the local health centre.
  Interventions: Behavioral: conventional community interventions

INTERVENTIONS:
Behavioral: prevention and management of childhood illnesses at community level — provision of critical health education and targeted promotion services to the participants in their locality
  Arms: Intervention arm
Behavioral: conventional community interventions — community health programs as the sole source of health education
  Arms: Conventional Intervention arm

SUMMARY:
This study modified and contextualized a community mobilization approach in a bid to find a solution to reduce the high incidence and prevalence of child morbidity and mortality in Zimbabwe.The developed model will be tested for its effectiveness in reducing child morbidity and mortality at community level by comparing the effect of the intervention to that of the conventional community interventions.

DETAILED DESCRIPTION:
In Zimbabwe the Neonatal and infant mortality rate are 31/1000 and 57/1000 respectively (ZDHS, 2011). Seventy -four percent of these death occur at community level due to the delay in deciding to seek care . The government of Zimbabwe has intensified facility based health systems though very little has been done in community health system strengthening yet there is glaring evidence from recent studies that the burden of infant and child morbidity and mortality is largely at community level. The effect of social mobilization approaches in reducing socio-cultural causes of morbidity and mortality is not known. Evidence base for participatory models and their effectiveness remains scanty and in-country, there is no approved , integrated community mobilization model that achieves saturation coverage in addressing all facets of community maternal newborn and child health along the continuum of care. Community immersion with health services is in line with the Alma Ata Declaration of the Primary Health Care approach that seeks to decentralize health services to the marginalized people. The study will test the effectiveness of the contextualized model in improving child health outcomes.

A cluster randomized controlled design will be used in 2 randomly selected districts of Mashonaland East , Zimbabwe. Women 18- 49 years with children 0-48 months in the selected districts will be recruited and followed up for 9-12 months . Stratified randomization will be used to select 11 pairs of participating villages . Central randomization will be employed for allocation concealment . The sample size was calculated in STATA 13. assuming a morbidity prevalence of 50% with a margin error of 5%. The assumed intra-cluster correlation coefficient (ICC) of 0.05 with a level of significance of 5% , design effect of 2.45 and power of 0.9. The sample size per arm will be 330 mother-child pairs and each arm will have 11 clusters.

Data will be collected monthly using monthly data collection tools. The study will require participants to commit at most 2 hours once in every two weeks. The main intervention is provision of critical health education and targeted promotion services to the participants in their locality. Participatory approaches will be employed in the intervention arm for learning and sharing of good community IMNCI practices for the prevention and management of childhood illnesses. Participants will be motivated through learning exchange visits and provision of promotional materials as incentives for successful completion and practice of recommended behaviors and child care practices.

ELIGIBILITY:
Inclusion Criteria:

Pregnant and lactating women staying in the study area with children below 4 years

Exclusion Criteria:

1. Women of child bearing age who do not dwell permanently in the study area
2. Women who are very ill and mentally challenged

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 765 (Actual)
Dates: Start 2017-01-19 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Reduction in child morbidity | 9- 12 months
  Incidence of childhood illnesses

SECONDARY OUTCOMES:
Early ANC uptake | 3 Months
  Number of women who booked in the first trimester
Institutional deliveries | 3 months
  Proportion of women with children 0-48 months who delivered at a health facility
Postnatal care uptake | 3 months
  Proportion of women with a child 0 -48 months who received post-natal care in their last delivery
Knowledge levels on child care | 3 months
  Proportion of women with a child 0-48 months who have basic knowledge on dangers signs and management of childhood illnesses

CONTACTS AND LOCATIONS:
Locations (1):
- College of Health Sciences, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Undecided